CLINICAL TRIAL: NCT01512849
Title: An Open-Label, Randomized, 2 Way Crossover, Single-Dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety of TA-7284 in Patients With Type 2 Diabetes Mellitus Who Have Moderate Renal Impairment
Brief Title: A Study to Evaluate the PK/PD and Safety of TA-7284 in Patients With Type 2 Diabetes Mellitus Who Have Moderate Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TA-7284-07
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: TA-7284; JNJ-28431754; Canagliflozin; Renal Impairment; Sodium Glucose Co-transporter2 (SGLT2) inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TA-7284 Low (Experimental)
  Interventions: Drug: TA-7284 Low
- TA-7284 High (Experimental)
  Interventions: Drug: TA-7284 High

INTERVENTIONS:
Drug: TA-7284 Low — Low
  Arms: TA-7284 Low
Drug: TA-7284 High — High
  Arms: TA-7284 High

SUMMARY:
The purpose of this study is to evaluate the PK/PD and safety of TA-7284 in patients with type 2 diabetes mellitus who have moderate renal impairment.

DETAILED DESCRIPTION:
This is an open-label, randomized, 2-way crossover study to evaluate the PK/PD and safety of TA-7284 in patients with type 2 diabetes mellitus who have moderate renal impairment relative to patients with type 2 diabetes mellitus who have normal renal function. The patients will receive both TA-7284-Low and TA-7284-High orally alone in either Period 1 or 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus in stable condition who have normal renal function or moderate renal impairment
* Body mass index of ≥18.5 kg/m2 and ≤39.9 kg/m2 at screening
* HbA1c of ≥6.5% and ≤10.5% at screening

Exclusion Criteria:

* Type 1 diabetes mellitus, diabetes mellitus resulting from pancreatic disorder, secondary diabetes mellitus
* Past or current history of severe diabetic complications
* Patients requiring insulin therapy
* History of hereditary glucose-galactose malabsorption or primary renal glucosuria

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nobuya Inagaki, MD, Study Director — Kyoto University, Graduate School of Medicine; Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation
Locations (1):
- Reserch site, Kanto, Japan

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818

RESULTS

PARTICIPANT FLOW:
Groups:
- Moderate Renal Impairment Low Dose First; Normal Renal Function Low Dose First: TA-7284 Low dose in Period 1, then crossover to TA-7284 High dose in Period 2
- Moderate Renal Impairment High Dose First; Normal Renal Function High Dose First: TA-7284 High dose in Period 1, then crossover to TA-7284 Low dose in Period 2
Period: Crossover Period 1
Arm/Group | Moderate Renal Impairment Low Dose First | Moderate Renal Impairment High Dose First | Normal Renal Function Low Dose First | Normal Renal Function High Dose First
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Crossover Period 2
Arm/Group | Moderate Renal Impairment Low Dose First | Moderate Renal Impairment High Dose First | Normal Renal Function Low Dose First | Normal Renal Function High Dose First
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Entire Population for Moderate Renal Impairment | Entire Population for Normal Renal Function | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Full Range); unit: years] | 63.7 (10.2) [40 to 78] | 57.8 (9.7) [48 to 76] | 60.8 [40 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Effect of Renal Function on Maximum Plasma Concentration of TA-7284
Time Frame: For 72 hours after each administration
Measure: Mean (Standard Deviation); unit: ng / mL
Groups:
- Moderate Renal Impairment Low; Normal Renal Function Low: TA-7284-Low was administered in a single dose.
- Moderate Renal Impairment High; Normal Renal Function High: TA-7284-High was administered in a single dose.
Arm/Group | Moderate Renal Impairment Low | Moderate Renal Impairment High | Normal Renal Function Low | Normal Renal Function High
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng / mL | 1197.1264 (310.5625) | 2333.3617 (414.8957) | 1213.6571 (337.8705) | 2415.6109 (739.8783)

2. Secondary Outcome: Adverse Events
Description: Incidence and severity of AEs
Time Frame: Upto approximately 14 days after last administration
Reporting Status: Not Posted

3. Secondary Outcome: 12-lead Electrocardiogram (ECG)
Description: Change from baseline in ECG parameters
Time Frame: For 72 hours after each administration
Reporting Status: Not Posted

4. Secondary Outcome: Vital Signs
Description: Change from baseline in Vital signs (BP, PR and BT)
Time Frame: For 72 hours after each administration
Reporting Status: Not Posted

5. Secondary Outcome: Clinical Laboratory Tests
Description: Change from baseline in Clinical laboratory tests
Time Frame: For 72 hours after each administration
Reporting Status: Not Posted

6. Primary Outcome: Effect of Renal Function on Area Under the Plasma Concentration-time Curve From Zero up to Infinity of TA-7284
Time Frame: For 72 hours after each administration
Measure: Mean (Standard Deviation); unit: ng･h/mL
Arm/Group | Moderate Renal Impairment Low | Moderate Renal Impairment High | Normal Renal Function Low | Normal Renal Function High
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng･h/mL | 8766 (2551) | 17835 (4434) | 6929 (1734) | 14815 (4162)

7. Primary Outcome: Effect of Renal Function on Urinary Glucose Excretion of TA-7284
Time Frame: For 24 hours after each administration
Measure: Mean (95% Confidence Interval); unit: g
Arm/Group | Moderate Renal Impairment Low | Moderate Renal Impairment High | Normal Renal Function Low | Normal Renal Function High
Number analyzed (Participants) | 12 | 12 | 12 | 12
g | 61.017 [49.362 to 72.671] | 70.904 [59.184 to 82.624] | 86.592 [75.612 to 97.572] | 103.052 [88.952 to 117.152]

8. Primary Outcome: Effect of Renal Function on Percent Inhibition of Renal Glucose Reabsorption (RGR) of TA-7284
Description: The percent inhibition of renal glucose reabsorption was calculated from renal glucose reabsorption (eGFR × plasma glucose AUC - urinary glucose excretion) on the preceding day and on the day of administration.
Time Frame: For 24 hours after each administration
Measure: Mean (95% Confidence Interval); unit: percent of RGR at baseline
Arm/Group | Moderate Renal Impairment Low | Moderate Renal Impairment High | Normal Renal Function Low | Normal Renal Function High
Number analyzed (Participants) | 12 | 12 | 12 | 12
percent of RGR at baseline | 60.8 [52.4 to 69.2] | 66.5 [59.5 to 73.5] | 47.8 [42.2 to 53.4] | 52.7 [45.4 to 60.0]

ADVERSE EVENTS:
Time Frame: Up to approximately 14 days after last administration
Description: Serious adverse events and the other adverse events were summarized in terms of renal function and dose.
Arm/Group | Moderate Renal Impairment Low | Moderate Renal Impairment High | Normal Renal Function Low | Normal Renal Function High
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/12 | 1/12 | 2/12 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate Renal Impairment Low (N=12) | Moderate Renal Impairment High (N=12) | Normal Renal Function Low (N=12) | Normal Renal Function High (N=12)
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 1
Blood creatin phosphokinase increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1
Protein urine present (Investigations) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other